CLINICAL TRIAL: NCT01764659
Title: Individually Optimized Contrast-Enhancement 4D-CT for Pancreatic Adenocarcinoma in Radiotherapy Simulation
Brief Title: 4D-CT for Pancreatic Adenocarcinoma in Radiotherapy Simulation
Acronym: GCC 1210
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Department of Radiation Oncology, Assistant Professor, Physics, University of Maryland, Baltimore
Other Study IDs: HP-00052534
Record Dates: First submitted 2013-01-02; First posted 2013-01-09 (Estimated); Results first posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: 4D-CT; Contrast Enhanced CT; Radiotherapy Simulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- All enrolled patients: Contrast-enhanced 4D computed tomography
  Interventions: Other: Contrast-enhanced 4D computed tomography

INTERVENTIONS:
Other: Contrast-enhanced 4D computed tomography — All enrolled patients each underwent three CT scans: a 4DCT immediately following a contrast-enhanced 3DCT and an individually optimized contrast-enhanced 4DCT.

SUMMARY:
The primary objective is to study the feasibility and efficacy of individually optimized CE 4D-CT for PDA in radiotherapy simulation.

DETAILED DESCRIPTION:
Compared with current clinical practice, the individually optimized CE 4D-CT can potentially provide much improved tumor-to-parenchyma conspicuity of pancreatic adenocarcinoma. This will help the radiation oncologists or radiologists to contour the tumor with higher precision and confidence, and compute the tumor volume and tumor motion more accurately.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years old or older
2. Patients with PDA who have not had surgical removal of their tumor and who are planned for treatment with radiotherapy in the Radiation Oncology Department at the University of Maryland.
3. Patients who have signed the contrast consent form and have been recommended by physicians to have contrast-enhanced CT scans.
4. Patients who have signed the consent form for this study

Exclusion Criteria:

1. Pregnant or breast-feeding women.
2. Patients with severely decreased renal function19-21.
3. Patients with known severe allergic reactions to contrast.
4. Patients who have difficulty lying flat on their back for extended periods of time.
5. Patients with breaths per minute (BPM) rate less than 10, due to the limitation of 4D-CT image reconstruction software.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: GI/GU multi-d clinic
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2013-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Lu, Ph. D., DABR, Principal Investigator — UMMC MSGCC; Hao H Zhang, Ph. D., Principal Investigator — UMMC
Locations (1):
- Ummc Msgcc, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Enrolled Patients: Individually optimized CE 4D-CT
Period: Overall Study
Arm/Group | All Enrolled Patients
Started | 14
Completed | 12
Not Completed | 2
Not completed — Death | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- GI Group: Study the feasibility and efficacy of individually optimized CE 4D-CT for PDA in radiotherapy simulation.
Arm/Group | GI Group
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Individually Optimized Contrast-enhanced 4DCT for Radiotherapy Simulation
Description: Image quality (anatomic details, motion artifacts, beam hardening and enhancement of pancreatic tissue and tumor were scored from 1 to 5, with 1 being very poor and 5 being excellent), CT number of pancreas and tumor, tumor-to-pancreas contrast, image noise and contrast-to-noise ration (CNR) were compared among contrast-enhanced (CE) 4DCT, CE 3DCT and 4DCT without contrast enhancement.
Time Frame: 1 year
Population: Image data of 10 patients (of the 12 patients who completed the study) was good for analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- CE 3DCT: Contrast-enhanced 3DCT
- 4DCT: 4DCT without contrast
- CE 4DCT: Individually optimized contrast-enhanced 4DCT
Arm/Group | CE 3DCT | 4DCT | CE 4DCT
Number analyzed (Participants) | 10 | 10 | 10
units on a scale
  Anatomic details | 4.1 (0.8) | 2.5 (0.6) | 3.6 (0.8)
  Motion artifacts | 3.9 (1.0) | 3.4 (0.9) | 3.7 (0.8)
  Beam hardening | 4.2 (0.8) | 3.3 (0.9) | 3.5 (0.8)
  Enhancement of pancreatic tissue and tumor | 3.2 (1.0) | 1.7 (0.9) | 3.3 (1.0)

2. Primary Outcome: Individually Optimized Contrast-enhanced 4DCT for Radiotherapy Simulation
Description: as for outcome 1
Time Frame: 1 year
Population: Image data of 10 patients (of the 12 patients who completed the study) was good for analysis.
Measure: Mean (Standard Deviation); unit: HU
Arm/Group | CE 3DCT | 4DCT | CE 4DCT
Number analyzed (Participants) | 10 | 10 | 10
HU
  Pancreas CT number (HU) | 49.2 (12.3) | 44.6 (15.9) | 75.5 (21.2)
  Tumor CT number (HU) | 53.0 (9.2) | 58.9 (14.3) | 76.3 (15.0)
  Tumor to pancreas contrast (HU) | 15.5 (20.7) | 9.2 (9.2) | 16.7 (12.3)
  Noise (HU) | 12.5 (3.9) | 19.4 (5.8) | 22.1 (5.7)

3. Primary Outcome: Individually Optimized Contrast-enhanced 4DCT for Radiotherapy Simulation
Description: as for outcome 1
Time Frame: 1 year
Population: Image data of 10 patients (of the 12 patients who completed the study) was good for analysis.
Measure: Mean (Standard Deviation); unit: contrast to noise ratio
Arm/Group | CE 3DCT | 4DCT | CE 4DCT
Number analyzed (Participants) | 10 | 10 | 10
contrast to noise ratio | 1.4 (1.9) | 0.6 (0.7) | 0.8 (0.6)

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- All Enrolled Patients: One death among enrolled patients, which was not directly related to this research.
Arm/Group | All Enrolled Patients
All-Cause Mortality (participants affected / at risk) | 1/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes